CLINICAL TRIAL: NCT04657484
Title: Comparison of the Efficacy and Safety of Two Corticosteroid Regimens in the Treatment of Diffuse Lung Disease After Coronavirus Disease 2019 (COVID-19) Pneumonia
Brief Title: Comparison of Two Corticosteroid Regimens for Post COVID-19 Diffuse Lung Disease
Acronym: COLDSTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2020/SPL-1528
Record Dates: First submitted 2020-12-05; First posted 2020-12-08 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Post COVID-19 Diffuse Lung Disease
Keywords: diffuse parenchymal lung disease; interstitial lung disease; organizing pneumonia; coronavirus disease-2019; SARS-Co-V-2
MeSH Terms: conditions — Lung Diseases, Interstitial; Organizing Pneumonia | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium dose prednisolone (Active Comparator): An initial dose of 40 mg/day will be administered for 1 week, followed by 30 mg/day for 1 week, 20 mg/day for 2 weeks, 10 mg/day for 2 weeks
  Interventions: Drug: Medium dose prednisolone
- Low dose prednisolone (Active Comparator): A dose of 10 mg/day of prednisolone will be administered for 6 weeks
  Interventions: Drug: Low dose prednisolone

INTERVENTIONS:
Drug: Medium dose prednisolone — Same as arm description
  Arms: Medium dose prednisolone
Drug: Low dose prednisolone — Same as arm description
  Arms: Low dose prednisolone

SUMMARY:
A proportion of patients with COVID-19 pneumonia have a prolonged course of illness. Some of these patients continue to have considerable respiratory symptoms or persistent hypoxemia. The CT abnormalities in these patients are often a combination of ground-glass opacities and patchy multifocal consolidation consistent with a pattern of OP. In several patients, these radiologic abnormalities persist. As with other forms of OP, patients with post-COVID OP or post COVID diffuse lung disease (PC-DLD) may benefit from treatment with oral glucocorticoids. The ideal dose of glucocorticoids for treating PC-DLD is unknown.

In this study, the investigatros aim to compare the efficacy and safety of a medium dose and a low dose of prednisolone (as the initial dose) for the treatment of post-COVID. diffuse lung disease.

DETAILED DESCRIPTION:
A proportion of patients with COVID-19 pneumonia (with or without ARDS) have a prolonged course of illness. Some of these patients continue to have considerable respiratory symptoms or persistent hypoxemia. The CT abnormalities in these patients are often a combination of ground-glass opacities and patchy multifocal consolidation consistent with a pattern of OP. In several patients, these radiologic abnormalities persist even after the symptoms of active COVID-19 have subsided and swabs from the upper respiratory tract for SARS-CoV-2 have turned negative. Such patients may be classified as having a secondary form of OP, namely post-infectious OP. Some of the patients also start developing signs of fibrosis.

As with other forms of OP, patients with post-COVID OP or post COVID diffuse lung disease (PC-DLD) may benefit from treatment with oral glucocorticoids.

Glucocorticoids may be a double-edged sword in this clinical situation. Steroids reduce inflammation associated with OP with a resultant resolution of symptoms, improvement in gas exchange (resulting in the resolution of hypoxemia), and potentially preventing the progression of early parenchymal abnormalities to irreversible fibrosis. However, they are associated with adverse effects such as hyperglycemia, delayed viral clearance, and increased susceptibility to infections. The ideal dose of glucocorticoids for treating PC-DLD is unknown. As PC-DLD is likely to get recognised early (much earlier than the average duration between onset of symptoms and diagnosis in other forms of OP, i.e., about 3-6 months), there is a possibility a lower intensity of glucocorticoids may be sufficient for treatment than the usual regimens, with the advantage of lesser adverse effects. A previous retrospective study that compared two regimens (higher dose intensity [DI] of glucocorticoids alone vs. glucocorticoids at a lower dose intensity along with clarithromycin), however, found that a complete radiologic response was higher in the prednisone alone (higher DI) group (81% vs. 63%) than in the combination group (with a lower DI of prednisone). Statistical significance was however not achieved (p=0.38), mainly due to the small sample size.

The investiagtors hypothesize that in PC-DLD a higher intensity (i.e., starting with a medium dose of prednisolone) will be more effective than a lower dose intensity (i.e., starting with a low dose of prednisolone) of glucocorticoids in effecting a radiologic response at six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed to have COVID-19 by means of a real-time reverse transcription polymerase chain reaction (rRT-PCR) test performed on a respiratory (upper or lower respiratory) sample or the detection of COVID-19 antigen
* Having significant respiratory symptoms (cough and breathlessness) or persistent hypoxemia or oxygen desaturation on exercise and CT chest showing residual changes of post-COVID parenchymal involvement of any extent OR having CT chest showing residual changes of post-COVID parenchymal involvement >20% of the lung parenchyma on visual inspection of the scans between 3-8 weeks of the onset of symptoms of COVID-19
* Willing to participate in the study

Exclusion Criteria:

* Receiving ventilatory or respiratory support (invasive or non-invasive mechanical ventilation or high flow nasal cannula) or supplemental oxygen with FiO2>0.35
* Requiring intensive care due to acute COVID-19 pneumonia or its complications
* Having a known lung parenchymal lung disease before the onset of COVID-19
* Pregnant or lactating women
* Having absolute contraindication for prednisolone in a dose of 40 mg/day (this includes untreated glaucoma, uncontrolled diabetes mellitus, signs of an uncontrolled or untreated infection or sepsis, pulmonary mycosis, untreated severe psychiatric disorders)
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a complete radiologic response | 6 weeks
  Complete response is defined as complete disappearance or ≥90% reduction in the lung parenchymal abnormalities on a high-resolution CT scan

SECONDARY OUTCOMES:
Proportion of subjects with a complete or good response radiologic response | 6 weeks
  Complete response is defined as complete disappearance or ≥90% reduction in the lung parenchymal abnormalities on a high-resolution CT scan. Good response is defined as ≥50% but less than 90% reduction in the lung parenchymal abnormalities on a high-resolution CT scan.
Proportion of subjects with a good composite response | 6 weeks
  Complete or good radiologic resolution along with no oxygen desturation on exercise testing and a normal spirometry
Forced vital capacity as a percentage of the predicted | 6 weeks
  Forced vital capacity will be measured using spirometry. The predicted value will be calculated based on standard reference equations.
Change in resting oxygen saturation | 6 weeks
  The change in resting oxygen saturation (measured by pulse oximetry) from the day of randomization to 6 weeks
Proportion of subjects with oxygen desaturation on exercise testing | 6 weeks
  Oxygen desaturation will be defined as a fall in oxygen saturation by 4% or more on exercise testing (by one-minute sit-to-stand test and six-minute walk test)
Change in dyspnea score on modified Medical Research Council scale | 6 weeks
  The change in dyspnea score assessed using the modified Medical Research Council from the day of randomization to 6 weeks.The scale has a minimum score of 0 and a maximum score of 4, higher values indicate worse outcomes
Severity of dyspnea on the Functional Assessment of Chronic Illness Therapy - Dyspnea-10 item scale | 6 weeks
  Severity of dyspnea assessed using the Functional Assessment of Chronic Illness Therapy - Dyspnea-10 item scale. The scale has two item banks of 10 items each for dyspnea and functional limitations. EAch item has a minimum score of 0 and maximum score of 3. Higher scores represent worse outcomes.
Change in respiratory health status using the King's Brief ILD questionnaire | 6 weeks
  Respiratory health status assessed using the King's Brief ILD questionnaire. The questionnaire has 15 items. The total score varies from 0 to 100, with higher scores representing better outcomes.
Change in health-related quality of life using the Short Form-36 questionnaire | 6 weeks
  Health-related quality of life assessed using Short Form-36 questionnaire. The questionnaire consists of 36 items covering 8 domains. Each domain score has a minimum value of 0 and maximum value of 100, with higher scores representing better outcomes
Proportion of subjects who develop adverse effects of prednisolone | 6 weeks
  The adverse effects of treatment (acne, weight gain, hyperglycemia, hypertension, abdominal pain, dyspepsia, Cushingoid facies, skin thinning and bruising, mood changes, muscular weakness and any other adverse effects related to prednisolone)

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhooria S, Chaudhary S, Sehgal IS, Agarwal R, Arora S, Garg M, Prabhakar N, Puri GD, Bhalla A, Suri V, Yaddanapudi LN, Muthu V, Prasad KT, Aggarwal AN. High-dose versus low-dose prednisolone in symptomatic patients with post-COVID-19 diffuse parenchymal lung abnormalities: an open-label, randomised trial (the COLDSTER trial). Eur Respir J. 2022 Feb 17;59(2):2102930. doi: 10.1183/13993003.02930-2021. Print 2022 Feb. PMID 34887325